CLINICAL TRIAL: NCT01632371
Title: ISAR-DESIRE 4: Randomized Trial Of Scoring Balloon in Patients With Restenosis in "Limus"-Eluting Coronary Stents Undergoing Angioplasty With Paclitaxel-Coated Balloon
Brief Title: Intracoronary Stenting and Angiographic Results: Optimizing Treatment of Drug Eluting Stent In-Stent Restenosis 4
Acronym: ISAR-DESIRE 4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE NO. S00112; CIV-12-05-006401 (Other: European Databank on Medical Devices (EUDAMED))
Record Dates: First submitted 2012-06-26; First posted 2012-07-02 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Restenosis; Stable Angina Pectoris; Acute Coronary Syndrome
Keywords: In-stent Restenosis; Drug Eluting Stent; Paclitaxel Coated Balloon; Scoring Balloon; Cutting Balloon; Angiographic follow-up; Optical coherence tomography (OCT)
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel Eluting Balloon + Scoring Balloon (Experimental): Dilatation of the lesion with an Paclitaxel Eluting Balloon before the utilization of a Scoring Balloon
  Interventions: Device: Paclitaxel Eluting Balloon + Scoring Balloon
- Paclitaxel Eluting Balloon (Active Comparator): Paclitaxel Eluting Balloon
  Interventions: Device: Paclitaxel Eluting Balloon

INTERVENTIONS:
Device: Paclitaxel Eluting Balloon + Scoring Balloon — Scoring/cutting balloon lesion predilation; paclitaxel eluting balloon therapy
  Arms: Paclitaxel Eluting Balloon + Scoring Balloon
Device: Paclitaxel Eluting Balloon — Standard balloon lesion predilation; paclitaxel-eluting balloon therapy
  Arms: Paclitaxel Eluting Balloon

SUMMARY:
The purpose of the study is to determine whether scoring balloon (SCB) plus paclitaxel-coated balloon (PCB) is superior to PCB alone for the treatment of restenosis within "limus"-eluting stents (LES)

DETAILED DESCRIPTION:
The optimal treatment of in-BMS-restenosis seems to be implantation of a DES which is supported by a large body of evidence. Nevertheless, several recent published studies have shown a substantial reduction in late lumen loss and angiographic restenosis using paclitaxel-coated balloons (PCB) for restenotic lesions. Given the increased world-wide use of DES and the use of DES in increasingly complex coronary disease patterns, the number of patients presenting with restenosis after DES implantation will further increase in the coming decade.

Data regarding the optimal treatment of in-DES-restenosis are very limited: Implanting a new DES for in-DES-restenosis has been reported to associate with repeat restenosis rates as high as 20%. In addition, an increased risk of stent thrombosis has been associated with complex stenting and with additional DES implantation. Thus, for lesions which develop restenosis after LES implantation, the optimal treatment strategy remains unknown.

Few results on small sample-size populations have been reported in patients treated with scoring or cutting balloon (SCB) technology for treatment of BMS restenosis as compared to plain balloon angioplasty. Moreover, the efficacy of SCB angioplasty in DES restenosis has not been adequately addressed. Furthermore, the potential additive benefit of SCB angioplasty in patients undergoing PCB therapy remains to be elucidated. The hypothesis behind this concept is that the application of SCB prior to deployment of PCB may increase the bioavailability of paclitaxel within the restenotic tissue, and therefore may increase the efficacy of PCB. There are numerous preclinical studies to support this hypothesis, which show that lesion preparation is an important pre-requisite for the effectiveness of PCB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% restenosis after prior implantation of LES in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

* Age < 18 years
* Cardiogenic shock
* Acute ST-elevation myocardial infarction within 48 hours from symptom onset.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Severe renal insufficiency (glomerular filtration rate ≤ 30 ml/min)
* Contraindications to antiplatelet therapy, paclitaxel, stainless steel, cobalt, chrome
* Therapy including Lovastatin, Ciclosporin, Terfenadine, Midazolam, or Ondansetron
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
In-segment percent diameter stenosis | 6-8 months
  In-segment percent diameter stenosis (%DS) at 6-8 month follow-up angiography

SECONDARY OUTCOMES:
In-stent late lumen loss | 6-8 months
  The difference between minimal lumen diameter post-procedure and minimal lumen diameter at follow-up angiography
In-segment binary angiographic restenosis | 6-8 month
  diameter stenosis ≥50% in the in-segment area (including the interventional area as well as 5 mm margins proximal and distal) at follow-up angiography
Death or myocardial infarction | 1 and 2 years
  Combined incidence of death or myocardial infarction at one and two year
Target lesion revascularization | 1 and 2 years
  Need for target lesion revascularization (TLR), defined as any revascularization procedure involving the target lesion due to luminal re-narrowing in the presence of symptoms or objective signs of ischemia at one and two year follow-up
Target lesion thrombosis | 1 and 2 years
  Incidence of target lesion thrombosis at one and two years
OCT tissue characterization | 6-8 months
  Tissue characterization following application of SCB and PCB using OCT at 6 -8 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Munich; Robert Byrne, MB PhD, Principal Investigator — Deutsches Herzzentrum Munich
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - 1. Med. Klinik am Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria

REFERENCES:
- [Derived] Kufner S, Joner M, Schneider S, Tolg R, Zrenner B, Repp J, Starkmann A, Xhepa E, Ibrahim T, Cassese S, Fusaro M, Ott I, Hengstenberg C, Schunkert H, Abdel-Wahab M, Laugwitz KL, Kastrati A, Byrne RA; ISAR-DESIRE 4 Investigators. Neointimal Modification With Scoring Balloon and Efficacy of Drug-Coated Balloon Therapy in Patients With Restenosis in Drug-Eluting Coronary Stents: A Randomized Controlled Trial. JACC Cardiovasc Interv. 2017 Jul 10;10(13):1332-1340. doi: 10.1016/j.jcin.2017.04.024. PMID 28683939